CLINICAL TRIAL: NCT05673980
Title: A Randomized Controlled Clinical Trial of Oral Vitamin D2 for the Prevention of COVID-19
Brief Title: Oral Vitamin D2 for Prevention of COVID-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Collaborators: Beijing Haidian Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: M2022828
Record Dates: First submitted 2022-12-30; First posted 2023-01-06 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2022-12

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Ergocalciferols; Cholecalciferol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vitamin D2 (Experimental): Oral dose of Vitamin D2 every two weeks
  Interventions: Drug: Vitamin D2
- Placebo (Placebo Comparator): Without any intervention
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Vitamin D2 — Participants in the vitamin D2 group received 200,000 IU of vitamin D2 orally on the first day of the trial and again two weeks later
  Other Names: cholecalciferol
  Arms: vitamin D2
Other: placebo — This group will not do any intervention
  Arms: Placebo

SUMMARY:
A total of 218 participants will be included in this study, and will be randomly assigned 1:1 to the group taking vitamin D2 and the group not taking vitamin D2. Participants in the group taking vitamin D2 orally will receive 200,000 IU of vitamin D2 on the first day of the trial, and again two weeks later (200,000 IU) . The group that will not receive vitamin D2 will not receive any intervention. The whole trial will laste four weeks.

DETAILED DESCRIPTION:
This study is a randomized controlled multicenter clinical trial. Participants who meet the inclusion criteria can be included in this trial after signing informed consent. A total of 218 participants will be included in this study, and will be randomly assigned 1:1 to the group taking vitamin D2 and the group not taking vitamin D2. Participants in the group taking vitamin D2 orally will receive 200,000 IU of vitamin D2 on the first day of the trial, and again two weeks later (200,000 IU) . The group that will not receive vitamin D2 will not receive any intervention. The whole trial will laste four weeks. Throughout the trial, participants' nucleic acid or antigen results, 25(OH)D concentrations, etc., need to be tested.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to participate in the clinical study and sign the informed consent;
2. Staff members of Peking University Third Hospital, including the hospital headquarters, Capital International Airport Hospital, North Hospital, Beijing Haidian Hospital, Peking University Third Hospital Yanqing Hospital and Peking University Third Hospital Chongli Hospital;
3. Test negative for COVID-19 antigen and have no symptoms related to COVID-19.

Exclusion Criteria:

1. Hospital staff with serious underlying diseases;
2. Pregnant and lactating women;
3. Long-term vegetarians;
4. Long-term chronic diarrhea, history of subtotal gastrectomy, biliary obstructive disease and pancreatic disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 218 (Estimated)
Dates: Start 2022-12-18 (Actual); Primary Completion 2023-01-19 (Estimated); Study Completion 2023-02-20 (Estimated)

PRIMARY OUTCOMES:
Change in incidence of laboratory-confirmed (or COVID-19 antibody test) COVID-19 infection | 4 weeks
  The test will be nucleic acid or antigen testing twice a week for four weeks

SECONDARY OUTCOMES:
The duration of a positive to negative antigen test after infection with COVID-19 | up to 4 weeks
  Antigen test results were recorded twice a week for four weeks
The duration of symptoms in COVID-19 positive participants | up to 4 weeks
  For COVID-19 positive participants, symptoms will be recorded on a questionnaire twice a week.
The proportion of participants whose symptoms of COVID-19 infection were confirmed by antigen testing for more than 7 days | 4 weeks
  For COVID-19 positive participants, symptoms will be recorded on a questionnaire twice a week.
The proportion of asymptomatic COVID-19 infected persons (those who test positive for the etiology of COVID-19 but have no related clinical manifestations) | 4 weeks
  For COVID-19 positive participants, symptoms will be recorded on a questionnaire twice a week.

CONTACTS AND LOCATIONS:
Overall Officials: Chunli Song, Pro., Study Chair — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Wang H, Liu H, Huang J, Meng X, Wang W, Xiao W, Liu D, Tao L, Song C. Comparative Effects of Minodronate and Alendronate on Low Back Pain in Postmenopausal Osteoporosis and Age Influence: A Head-to-Head, Randomized Clinical Trial. Clin Interv Aging. 2025 Nov 27;20:2219-2230. doi: 10.2147/CIA.S541940. eCollection 2025. PMID 41341143
- [Derived] Wang H, Tao L, Cui L, Chen Y, Liu D, Xue L, Yang Y, Lv Y, Zhang F, Wang T, Wang X, Yuan W, Liu H, Huang J, Jiang Y, Liu N, Yang L, Hu Y, Li Y, Gao Y, Li H, Li B, Song C. Randomized trial of influence of vitamin D on the prevention and improvement of symptomatic COVID-19. Sci Rep. 2024 Sep 3;14(1):20519. doi: 10.1038/s41598-024-66267-8. PMID 39227626